CLINICAL TRIAL: NCT06350097
Title: A Phase III, Open-label, Randomised Study of Osimertinib With or Without Datopotamab Deruxtecan (Dato-DXd), as First-line Treatment in Participants With Epidermal Growth Factor Receptor (EGFR) Mutation-positive, Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Phase III, Open-label Study of First-line Osimertinib With or Without Datopotamab Deruxtecan for EGFRm Locally Advanced or Metastatic Non-small Cell Lung Cancer
Acronym: TROPION-Lung14
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D516NC00001; 2023-509883-89-00 (Other: EU CT Number)
Record Dates: First submitted 2024-04-02; First posted 2024-04-05 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer, NSCLC, Epidermal Growth Factor Receptor (EGFR) Mutation-positive, Osimertinib, Dato-DXd, Datopotamab Deruxtecan, Tagrisso
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Osimertinib in combination with Datopotamab Deruxtecan (Experimental): Participants in this group will receive osimertinib 80 mg QD as oral tablet with Datopotamab Deruxtecan 6mg/kg as i.v. infusion q3w of Day 1 of every 21-day cycle.
  Interventions: Drug: Osimertinib; Drug: Datopotamab Deruxtecan
- Arm 2: Osimertinib monotherapy (Active Comparator): Participants in this group will receive osimertinib 80 mg QD as oral tablet.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Arm 1: Osimertinib 80 mg QD as oral tablet with Datopotamab Deruxtecan 6mg/kg as i.v. infusion.
  Arm 2: Osimertinib 80 mg QD as oral tablet .
  Other Names: Osimertinib: AZD9291
Drug: Datopotamab Deruxtecan — Osimertinib 80 mg QD as oral tablet with Datopotamab Deruxtecan 6mg/kg as i.v. infusion.
  Other Names: Datopotamab Deruxtecan: Dato-DXd, DS-1062a
  Arms: Arm 1: Osimertinib in combination with Datopotamab Deruxtecan

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of osimertinib (tablet) in combination with Dato-DXd (i.v. infusion) compared with osimertinib (tablet) monotherapyas a first-line therapy in participants with locally advanced or metastatic EGFRm (Ex19del and/or L858R) NSCLC.

Study details include:

1. The study duration will be event-driven, with an estimated duration of approximately 9 years.
2. Participants may receive study treatment until disease progression, unacceptable toxicity, or other specific discontinuation criteria are met.
3. The visit frequency will be every 3 weeks during the treatment period.

Note: Participants on osimertinib treatment(osimertinib only arm or who have discontinued Dato-DXd while are still receiving osimertinib) are required to attend visits to perform assessments every 6 weeks from Cycle 7 until Cycle 17 and then visits every 12 weeks until disease progression or IP discontinuation. Participants who are receiving osimertinib + Dato-DXd are still required to attend visit to perform assessment every 3 weeks (q3w) per SoA.

DETAILED DESCRIPTION:
This is a global Phase III, open-label, randomised, multicentre study assessing the efficacy and safety of osimertinib in combination with Datopotamab Deruxtecan compared with osimertinib in participants with locally advanced or metastatic EGFRm (Ex19del and/or L858R) NSCLC who have not received any prior therapy for advanced disease.

ELIGIBILITY:
Inclusion Criteria:

Age

1. Participant must be ≥ 18 years.

   Type of Participant and Disease Characteristics
2. Histologically or cytologically documented nonsquamous NSCLC. NSCLC of mixed histology is allowed if adenocarcinoma is the predominant histology. Mixed small-cell lung cancer and NSCLC histology, and sarcomatoid variant of NSCLC is ineligible.
3. Stage IIIB or IIIC or Stage IV metastatic NSCLC or recurrent NSCLC (based on the American Joint Committee on Cancer Edition 8) not amenable to curative surgery or definitive chemoradiation at the time of randomisation.
4. Participants must not have received prior EGFR TKIs or other systemic therapy for Stage IIIB, IIIC or IV NSCLC.
5. The tumour harbors at least 1 of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del or L858R), either alone or in combination with other genomic alterations, which may include EGFR T790M, assessed by a CLIA-certified (US sites) or an accredited (outside of the US) local laboratory or by central prospective tissue testing.
6. For participants enrolled in randomisation period, mandatory provision of an unstained, archival tumour tissue sample in a quantity sufficient to allow for central confirmation of the EGFR mutation status.
7. WHO performance status of 0 or 1.
8. At least one lesion not previously irradiated that qualifies as a RECIST 1.1 TL at baseline and can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have short axis ≥15 mm) with CT or MRI and is suitable for accurate repeated measurements.
9. Adequate bone marrow reserve and organ function within 7 days before the first dose of study intervention.

   Sex and Contraceptive/Barrier Requirements
10. Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

    Other Inclusion Criteria
11. All races, gender and ethnic groups are eligible for this study.

Exclusion Criteria:

1. As judged by the investigator, any evidence of diseases (such as severe or uncontrolled systemic diseases, including active bleeding diseases, psychiatric illness/social situations), history of allogenic organ transplant, and/or substance abuse which, in the investigator's opinion, makes it undesirable for the participant to participate in the study or that would jeopardise compliance with the protocol.
2. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption, distribution, metabolism, or excretion of osimertinib.
3. History of another primary malignancy.
4. Spinal cord compression and unstable brain metastases, as defined by Protocol.
5. Clinically significant corneal disease.
6. Has active or uncontrolled hepatitis B or C virus infection, as defined by Protocol.
7. Known HIV infection that is not well controlled, as defined by Protocol.
8. Uncontrolled infection requiring i.v. antibiotics, antivirals or antifungals; suspected infections (eg, prodromal symptoms); or inability to rule out infections (participants with localised fungal infections of skin or nails are eligible).
9. Resting ECG with clinically abnormal findings, as defined by Protocol.
10. Uncontrolled or significant cardiac disease, as defined by Protocol.
11. Past medical history of ILD/penumonitis, including radiation pneumonitis (apart from radiation pneumonitis that did not require steroids), or drug-induced ILD/pneumonitis, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
12. Pulmonary embolism within 3 months of the study enrolment or has severe pulmonary function compromise.

    Prior/Concomitant Therapy
13. Prior exposure to any agent including an ADC containing a chemotherapeutic agent targeting topoisomerase I, TROP2-targeted therapy.

    Prior/Concurrent Clinical Study Experience
14. Participants with a known history of severe hypersensitivity reactions to either Dato-DXd and osimertinib or any excipients of Dato DXd and osimertinib or drugs with a similar chemical structure or class to DXd and osimertinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2028-03-21 (Estimated); Study Completion 2032-05-25 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the superiority of osimertinib in combination with Datopotamab Deruxtecan relative to osimertinib by assessment of Progression Free Survival (PFS) by BICR in all randomised participants. | It is anticipated that it will be performed approximately 3 years after the first participant is randomised.
  PFS is defined as time from randomisation until progression per RECIST 1.1 as assessed by BICR, or death due to any cause (in the absence of progression).

SECONDARY OUTCOMES:
To demonstrate the superiority of osimertinib in combination with Datopotamab Deruxtecan relative to osimertinib by assessment of Overall Survival (OS) in all randomised participants. | It is anticipated that it will be performed approximately 7 years after the first participant has been randomised.
  OS defined as the time from randomisation until the date of death due to any cause.
To demonstrate the effectiveness of osimertinib in combination with Datopotamab Deruxtecan relative to osimertinib by assessment of PFS on Central nervous system (CNS) metastases in participants with CNS metastases at baseline | It is anticipated that it will be performed approximately 3 years after the first participant is randomised.
  Central nervous system progression-free survival (CNS PFS) is defined as the time from randomisation until the date of objective CNS progression assessed by CNS BICR or death (by any cause in absence of CNS progression).
To demonstrate the effectiveness of osimertinib in combination with Datopotamab Deruxtecan relative to osimertinib by assessment of PFS by investigator in all randomised participants. | It is anticipated that it will be performed approximately 3 years after the first participant is randomised.
  PFS is defined as time from randomisation until progression per RECIST 1.1 as assessed by investigator, or death due to any cause (in the absence of progression).
To demonstrate the effectiveness of osimertinib in combination with Datopotamab Deruxtecan relative to osimertinib by assessment of Overall Response Rate (ORR) in all randomised participants with measurable disease at baseline. | It is anticipated that it will be performed approximately 3 years after the first participant is randomised.
  ORR is defined as the proportion of participants who have a confirmed Complete Response (CR) or confirmed Partial Response (PR), as determined by BICR (and investigator) per RECIST 1.1.
To demonstrate the effectiveness of osimertinib in combination with Datopotamab Deruxtecan relative to osimertinib by assessment of Duration of Response (DoR) in all randomised participants with measurable disease at baseline. | It is anticipated that it will be performed approximately 3 years after the first participant is randomised.
  DoR is defined as the time from the date of first documented confirmed response until date of documented progression per RECIST 1.1, as assessed by BICR (and investigator) assessment or death due to any cause.
  The measure of interest is the median of DoR.
To demonstrate the effectiveness of osimertinib in combination with Datopotamab Deruxtecan relative to osimertinib on the prevention of CNS metastases | It is anticipated that it will be performed approximately 3 years after the first participant is randomised.
  Neuro-radiologist assessments according to CNS RECIST 1.1 to determine the presence/absence of CNS lesions at progression in participants without CNS metastases at baseline.
To demonstrate the effectiveness of osimertinib in combination with Datopotamab Deruxtecan relative to osimertinib by assessment of PFS2 in all randomised participants | It is anticipated that it will be analyzed by time of PFS primary which is about 3 years after the first participant has been randomised.
  PFS2 will be defined as the time from randomisation to the earliest of the progression event (following the initial progression) subsequent to first subsequent anti-cancer therapy, or death.
To assess the Pharmacokinetics (PK) of osimertinib and Datopotamab Deruxtecan | It is anticipated that it will be performed approximately 3 years after the first participant has been randomised.
  Concentration of osimertinib and its metabolite AZ5104, Datopotamab Deruxtecan, total anti-TROP2 antibody and DXd in plasma.
To investigate the immunogenicity of Datopotamab Deruxtecan | It is anticipated that it will be performed approximately 3 years after the first participant has been randomised, together with PFS primary.
  Presence of ADAs for Datopotamab Deruxtecan (confirmatory results: positive or negative, titres, and neutralizing antibodies).
To compare the local EGFR mutation test result used for patient selection with the retrospective central cobas® EGFR Mutation Test v2 results from baseline tumour samples | It is anticipated that it will be performed approximately 3 years after the first participant is randomised.
  Concordance of EGFR mutation status between the local EGFR mutation test and the central cobas® EGFR Mutation Test v2 results from tumour samples with evaluable results.
To demonstrate the effectiveness of osimertinib in combination with Datopotamab Deruxtecan vs. osimertinib monotherapy based on the cobas® EGFR Mutation Test v2 plasma screening test result for Ex19del or L858R EGFR mutations | It is anticipated that it will be performed approximately 3 years after the first participant has been randomised, together with PFS primary.
  PFS by Investigator by plasma EGFR mutation status PFS is defined as time from randomisation until progression per RECIST 1.1 as assessed by investigator, or death due to any cause (in the absence of progression).

CONTACTS AND LOCATIONS:
Locations (141):
- United States (32):
  - Research Site, Fountain Valley, California
  - Research Site, Los Alamitos, California
  - Research Site, Los Angeles, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Santa Monica, California
  - Research Site, Walnut Creek, California
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Ocala, Florida
  - Research Site, Orange City, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, North Chicago, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Bethesda, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Saint Paul, Minnesota
  - Research Site, Bridgeton, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Brooklyn, New York
  - Research Site, New York, New York
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Webster, Texas
  - Research Site, Woodway, Texas
  - Research Site, Fairfax, Virginia
  - Research Site, Fort Belvoir, Virginia
  - Research Site, Midlothian, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Milwaukee, Wisconsin
- Australia (5):
  - Research Site, Camperdown
  - Research Site, Clayton
  - Research Site, Kogarah
  - Research Site, South Brisbane
  - Research Site, Westmead
- Brazil (5):
  - Research Site, Barretos
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Edmonton, Alberta
  - Research Site, Montreal, Quebec
- China (21):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Linhai
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Zhengzhou
- France (4):
  - Research Site, Angers
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Strasbourg
- Germany (9):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Erfurt
  - Research Site, Frankfurt
  - Research Site, Göttingen
  - Research Site, Immenhausen
  - Research Site, Kiel
  - Research Site, Mainz
  - Research Site, München
- Hong Kong (3):
  - Research Site, Hong Kong
  - Research Site, Jordan
  - Research Site, Lai Chi Kok
- India (10):
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Kolkata
  - Research Site, Mysuru
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Vadodara
  - Research Site, Varanasi
- Italy (5):
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Orbassano
  - Research Site, Padua
  - Research Site, Parma
- Japan (11):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Wakayama
  - Research Site, Yokohama
- Poland (4):
  - Research Site, Bystra
  - Research Site, Olsztyn
  - Research Site, Poznan
  - Research Site, Warsaw
- Puerto Rico (2):
  - Research Site, Rio Piedras
  - Research Site, San Juan
- South Korea (4):
  - Research Site, Erie
  - Research Site, Goyang-si
  - Research Site, Namdong-gu
  - Research Site, Seoul
- Spain (6):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Valencia
- Taiwan (4):
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Dusit
  - Research Site, Hat Yai
  - Research Site, Udon Thani
- Turkey (Türkiye) (6):
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Goztepe Istanbul
  - Research Site, Izmir
  - Research Site, Küçükçekmece
  - Research Site, Seyhan
- Vietnam (4):
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Vinh

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/